CLINICAL TRIAL: NCT00656331
Title: The Pleiotropic Effects of Atorvastatin When Combined With Common Antihypertenisve Medications: A Comparison of Amlodipine and Hydrochlorothiazide
Brief Title: The Pleiotropic Effects of Atorvastatin When Combined With Common Antihypertenisve Medications.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 05-106
Record Dates: First submitted 2008-04-07; First posted 2008-04-11 (Estimated); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Amlodipine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Amlodipine
  Interventions: Drug: Amlodipine and Hydrocholorothiazide
- 2 (Active Comparator): HCTZ
  Interventions: Drug: Amlodipine and Hydrocholorothiazide

INTERVENTIONS:
Drug: Amlodipine and Hydrocholorothiazide — Arm 1 gets Amlodipine and Arm 2 gets Hydrocholorothiazide

SUMMARY:
The purpose of this study is to compare the effects of the cholesterol medication taken with each blood pressure medication alone on heart disease risk factors including blood pressure, cholesterol, inflammation, blood sugar control, blood vessal function, and other heart disease risk factors.

ELIGIBILITY:
Inclusion Criteria:

* mild hypertension and high cholesterol

Exclusion Criteria:

* diabetes and heart disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-08; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
PAI-1 | study completion

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Colleran, MD, Principal Investigator — University of New Mexico
Locations (1):
- UNMHSC, Albuquerque, New Mexico, United States